CLINICAL TRIAL: NCT06685965
Title: A Phase-2, Double-Blind, Randomized, Placebo-controlled, Crossover Dose-Finding, Laboratory-based Study to Evaluate Effects on Sleep and Safety of RE03 in PTSD Patients With Sleep Disturbances
Brief Title: A Study to Evaluate Effects on Sleep and Safety of RE03 in PTSD Patients With Sleep Disturbances
Acronym: PTSD-PoC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reconnect Labs (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RL004
Record Dates: First submitted 2024-11-08; First posted 2024-11-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Sleep Disturbances and Insomnia
Keywords: Phase 2; Proof of Concept; Target Engagement; Cross-over; placebo-controlled; randomized; Sleep Disturbances; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Cross-over assignment: low dose, high dose and a placebo in randomized order
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): low dose of RE03
  Interventions: Drug: RE03
- High dose (Experimental): High dose of RE03
  Interventions: Drug: RE03
- Placebo control (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RE03 — Buccal Dexmedetomidine
  Arms: High dose; Low dose
Drug: Placebo — Matching Placebo
  Arms: Placebo control

SUMMARY:
Post-traumatic stress disorder (PTSD) affects many people who have experienced traumatic events. A common issue with PTSD is severe sleep disturbances, such as nightmares. Current treatments often do not provide sufficient relief, especially for sleep problems. This study aims to determine whether dexmedetomidine - a medication already used in intensive care - can improve sleep quality in PTSD patients.

DETAILED DESCRIPTION:
Participants spend one screening night followed by three treatment nights in the sleep lab, where they receive either a low dose, a high dose of dexmedetomidine, or a placebo. All participants receive all three options, with only the sequence differing. Participants and the study team are blinded and thus do not know which dose (or placebo) has been assigned.

ELIGIBILITY:
Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Male or female, aged ≥18 and ≤64 years (inclusive)
* Diagnosis of PTSD according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) for more than 6 months
* PTSD diagnosis assessed with CAPS-5 (life-time) severity ≥ 2
* Sleep disturbance, e.g., difficulty falling or staying asleep, or restless sleep (Criterion E6 of the DSM-5 criteria for PTSD) is present for at least a month prior to screening and causes clinically significant distress or impairment in social, occupational, or other important areas of functioning
* Sleep disturbance assessed with the PSQI; severity ≥ 5
* Ability (verified by investigator) and willingness to provide informed consent as documented by dated signature

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Inability to comply with sleep-wake schedule related study requirements, e.g. due to crossing of time zones (≥ 2), extreme chronotypes, shift working within 2 weeks prior to the screening visit, or planned shift work during the study, self-reported usual daytime napping ≥1 hour per day, and ≥3 days per week
* Inability to follow the procedures of the study, e.g. due to insufficient understanding of the German language used in the study as evaluated by the investigator or anticipated problems with overnight stays at the sleep laboratory
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dose; administration of a biological product (e.g. vaccines, blood components, gene therapies, tissues, etc.) in the context of a clinical research study within 90 days prior to the first dose; or concomitant participation in an investigational study involving drug or device administration
* Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomised at least 6 months prior to the first study drug administration) not willing to use one of the following acceptable contraceptive methods throughout the study and for at least 3 months after the last study drug administration:

  ○ Simultaneous use of condom and hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to sexual intercourse for the female partner;
* Females of non-childbearing potential who are neither:

  * Post-menopausal (status defined as an absence of menses for at least 12 months prior to the first study drug administration); or
  * Surgically sterilized (complete hysterectomy or bilateral oophorectomy at least 3 months prior to the first study drug administration)
* Male participants who are not vasectomised for at least 6 months prior to dosing and who are sexually active with a female partner of childbearing potential not willing to use one of the following acceptable contraceptive methods from the first dose and for 3 months after the last dose:

  ○ Use of condom and/or hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to sexual intercourse for the female partner;
* Male participants (including men who have had a vasectomy) with a pregnant partner not willing to use a condom from the first dose and for 3 months after the last dose.
* Male participants not willing to abstain from sperm donation for 3 months after the last dose
* Body Mass Index lower than 17.5 kg/m2 or higher than 35 kg/m2
* History of any clinically significant cardiovascular disorder, including:

  * Clinically significant atrioventricular conduction disturbance (e.g. higher grade AV block >grade 1), cardiac arrhythmias, sick sinus syndrome, or accessory bypass tract (e.g. Wolff-Parkinson-White)
  * Patients with symptomatic, or pronounced and persistent bradycardia (heart rate < 50 bpm) assessed during medical screening (during daytime)
  * Patients with persistent tachycardia (heart rate > 100 bpm) assessed during medical screening (during daytime)
  * Patients with hypotension (sBP < 90 mmHg, dBP < 50 mmHg), orthostatic dysregulation or a history of syncopes (e.g. micturition syncope)
  * Patients with hypertension ≥ Grade 2 (sBP ≥ 160 mmHg, dBP ≥ 100 mmHg)
  * Patients with a trend towards a baseline prolongation of the QT/QTc interval (men: >440 ms; women: >450 ms) at the screening visit, a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, hypomagnesemia, family history of Long QT syndrome)
  * Patients with history of myocardial infarction or coronary ischemia
  * Patients with cerebrovascular disease (e.g. Stroke, Hemorrhage, Transient Ischemic Attack, Aneurysm, Arteriovenous Malformation, Venous Thrombosis, Hematoma, etc.)
* Patients with peripheral arterial occlusive disease
* Patients with epilepsy, a history of seizures, or a history of severe head trauma or stroke
* Patients with chronic Obstructive Pulmonary Disease, pulmonary fibrotic disease or generally restrictive pulmonary disease, and related conditions which may cause respiratory depression under RE03 treatment
* Patients with any unstable medical condition, significant medical disorder or acute illness/injury (e.g. high fever) which, in the opinion of the Investigator, would jeopardize the safety of the participant, raise doubts about the feasibility of adhering to the trial protocol, or impact the validity of the study results
* Any laboratory test results deemed clinically significant by the Investigator, especially parameters relating to hepatic (Aspartate / Alanine aminotransferase) or renal metabolism / insufficiency (creatinine clearance) or diagnosed thyroid dysfunction (hypothyroidism or hyperthyroidism)
* Patients with abnormal liver function
* Suicidality (C-SSRS severity ≥ 4)
* Suicide attempt in the last 12 months
* Sleep-related conditions that may contribute to insomnia symptoms assessed via the Structured Clinical Interview for Sleep Disorders-Revised (SCISD-R) and PSG screening including:

  * Restless Leg Syndrome
  * Obstructive Sleep Apnea
  * Narcolepsy
  * Delayed-Sleep Phase Syndrome
  * REM Sleep Behaviour disorder
  * NREM Sleep Arousal disorder
* Prior or ongoing bipolar disorder, any psychotic disorder, including schizophrenia, schizophreniform disorder, schizoaffective disorder, brief psychotic disorder (unless substance induced or due to a medical condition), as assessed by a structured clinical interview (QuickSCID-5)
* Ongoing obsessive-compulsive disorder, or anorexia nervosa as assessed by medical history and a structured clinical interview (QuickSCID-5)
* Have a current moderate (not in early remission in the 3 months prior to enrollment; meets 5 of 11 diagnostic criteria per DSM-5) or severe alcohol use disorder within the 12 months prior to enrollment (meets at least 6 of 11 diagnostic criteria per DSM-5, QuickSCID-5)
* Current diagnosis of severe Substance-Use disorder (SUD) for nicotine (i.e. inability to refrain from smoking during the night) and cannabis (i.e. inability to refrain from smoking on study days) , and mild SUD for all other substances according to DSM-5 (QuickSCID-5)
* Concurrent daily and/or frequent use of any of the following restricted concomitant medications:

  * Inability or unwillingness to withdraw sedative medications for the duration of the study, including hypnotics, sedative antidepressants, sedative neuroleptics, antihistamines, dual orexin receptor antagonists (DORAs), agomelatine, melatonin, etc. for a minimum of 5 half-lives plus 1 week for stabilization (or at the discretion of the investigator) until the end of the study
  * Concomitant use of RE03 with beta-blockers, due to increased risk of bradycardia; currently unstable or recent changes in antihypertensive medication.
  * Unstable Antidepressant treatment initiated less than 3 months prior to screening
  * Concomitant use of RE03 with drugs with a risk for QT interval prolongation requires careful monitoring, in case clinically relevant QTc thresholds are exceeded during the trial (male > 470 ms; female > 480 ms), patients must be discontinued.
* Participants must not be currently enrolled in a psychological therapy program that involves varying frequency of sessions or different therapists throughout the study duration. Additionally, they should not have started any psychological therapy within 30 days prior to the screening or during the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Time spent in sleep stages N2 + N3 | 0.5 hours after each substance administration for 9 hours or until terminal morning awakening
  The total duration (in minutes) of sleep stages N2+N3, as measured by polysomnography (PSG) on the night following administration of each treatment [minutes spent in N2 + N3].

SECONDARY OUTCOMES:
REM fragmentation index | 0.5 hours after each substance administration for 9 hours or until terminal morning awakening
  The rapid eye movement (REM) fragmentation index as measured by polysomnography (PSG) on the night following administration of each treatment [# of entries from REM sleep into stage N1 or wake divided by total sleep time].

CONTACTS AND LOCATIONS:
Overall Officials: Andres Ort, MD, Principal Investigator — University of Zurich
Locations (1):
- Human Sleep Pharmacology, University of Zurich, Zurich, Canton of Zurich, Switzerland